CLINICAL TRIAL: NCT01455766
Title: Pulmonary Edema Following Major Thoracic Resections: a Value of Perioperative Volumetric Monitoring
Brief Title: Volumetric Monitoring in Major Lung Surgery
Acronym: EVLW-PNEUMO
Status: Completed | Type: Observational
Sponsor: Northern State Medical University (Other)
Collaborators: Regional hospital of Arkhangelsk (Unknown); University of Tromso (Other)
Responsible Party: Principal Investigator, Vsevolod V. Kuzkov, Associate Professor, MD, PhD, Northern State Medical University
Other Study IDs: 2005-2011
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Pneumonectomy; Acute Pulmonary Edema
Keywords: postpneumonectomy pulmonary edema; extravascular lung water

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma for non-specified additional retrospective tests.
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis of this observational single-center clinical study was to explore the volumetric hemodynamic monitoring in the perioperative period in major and risky thoracic intervention. The investigators monitored the changes in the volumes of blood in the central vessels and heart chambers as well as a volume of fluid in pulmonary tissue (i. e. extravascular lung water).

DETAILED DESCRIPTION:
The goal of this observational study is to investigate into changes in volumetric hemodynamic parameters obtained with a technique of transpulmonary indicator dilution after major thoracic intervention, including pneumonectomy and lobar resections. The important parameters of hemodynamics were monitored throughout the intervention and 48 hrs postoperatively, including extravascular lung water index, global end-diastolic volume index, etc.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age above 18 and below 80
* Confirmed malignant bronchial neoplasm or
* Destructive pulmonary infection

Exclusion Criteria:

* Pregnant
* Severe pulmonary hypertension
* Pulmonary tuberculosis
* Severe occlusive atherosclerosis of lower extremities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes the patients scheduled for extended thoracic resections (lobar resection and pneumonectomy) due to bronchial cancer or severe destructive pulmonary infection (abscess and/or pneumonia).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-02 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vsevolod V. Kuzkov, MD, PhD, Principal Investigator — Northern State Medical University; Mikhail M. Orlov, MD, Principal Investigator — Regional hospital of Arkhangelsk; Mikhail Y. Kirov, MD, PhD, Study Chair — Northern State Medical University; Lars J. Bjertnaes, MD, PhD, Study Director — University of Trmsoe, Tromsoe, Norway
Locations (1):
- Regional Hospital of Arkhangelsk, Arkhangelsk, Arkhangelskaya oblast, Russia